CLINICAL TRIAL: NCT03230422
Title: A Comparison of the Novel King Vision Pediatric aBlade and the C-MAC Video Laryngoscope to the Direct Laryngoscope in Simulated Normal and Difficult Infant Airway. A Bicentric, Prospective, Randomized Manikin Study
Brief Title: A Comparison of Video Laryngoscopes and the Direct Laryngoscope in Simulated Normal and Difficult Infant Airway.
Acronym: Kivi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Marc Kriege, MD, Dr. med. Marc Kriege, Dr. med. Nina Pirlich, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Johannes GU
Record Dates: First submitted 2017-07-23; First posted 2017-07-26 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Airway Complication of Anesthesia
Keywords: infant, laryngoscopes, pediatrics

STUDY DESIGN:
Who Masked: Participant
Masking Description: residents, fellows and attending with different level of experience
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- normal airway (Experimental): Time (normal airway) using the novel King Vision™ Pediatric aBlade (KV) video laryngoscope, C-MAC™ D-blade Ped (DP), C-MAC™ Miller Blade (MB), shortened as VL, compared with conventional direct laryngoscopy (DL)
  Interventions: Device: normal airway; Device: difficult airway
- difficult airway (Experimental): Time (difficult airway) using the novel King Vision™ Pediatric aBlade (KV) video laryngoscope, C-MAC™ D-blade Ped (DP), C-MAC™ Miller Blade (MB), shortened as VL, compared with conventional direct laryngoscopy (DL)
  Interventions: Device: normal airway; Device: difficult airway

INTERVENTIONS:
Device: normal airway — The Time interval between the laryngoscope blade passing the teeth/gums to the announcing of the first ventilation was recorded as the time to ventilation with the Video laryngoscopy (VL) or conventional direct laryngoscopy (DL)
Device: difficult airway — The Time interval between the laryngoscope blade passing the teeth/gums to the announcing of the first ventilation was recorded as the time to ventilation with the Video laryngoscopy (VL) or conventional direct laryngoscopy (DL)

SUMMARY:
In Pediatric both manikin and human studies have suggested that the video laryngoscopy is equally suitable to facilitate intubation compared to the direct laryngoscopy.

DETAILED DESCRIPTION:
The King Vision Pediatric aBlade is a novel video laryngoscopy for securing the airway of new born and infants. In this manikin studie we want to compare different types of video laryngoscopes in a simulated normal and difficult infant airway.

ELIGIBILITY:
Inclusion Criteria:

- anesthesiologists or neonatal/pediatric intensive care medicice specialists with experience in securing pediatric airway

Exclusion Criteria:

- participants without experience in pediatric airway management

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-09-27 (Actual)

PRIMARY OUTCOMES:
Time to ventilation (seconds) | Assessed intraoperatively at time of intubation (seconds)
  Three timepoints will be recorded, beginning with the insertion of the device past the theeth/gum into the mouth. These will inlcude time to best view, time to removal of device from the mouth, and the time to the first chest raising of the simulator

SECONDARY OUTCOMES:
First attempt success rate of tracheal intubation (in 40 seconds) | Assessed intraoperatively at time of intubation
  An attempt at tracheal intubation will be defined as entry of the device into the patient's mouth without the need to remove the device once entered and securing the airway.
Grades of Laryngeal View (Cormack&Lehane Class) | Assessed intraoperatively at time of intubation
  Cormack&Lehane Grade (1-4) and percentage of glottic opening (POGO) (%) will be recorded after insertion of the laryngoscope
Use of ELM | Assessed intraoperatively at time of intubation
  BURP or change the head/Shoulder position to optimised the glottic view will be recorded
Intubation Adjustments & Ease of Use | Assessed intraoperatively following intubation
  Airway manipulations utilized and ease of use (Likert 1-5) will be assessed by the user following the intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kriege, MD, Principal Investigator — University Medical Centre Mainz
Locations (1):
- Department of Anesthesiology,Prof. C. Werner, Universitätsmedizin of the JG University, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jagannathan N, Hajduk J, Sohn L, Huang A, Sawardekar A, Albers B, Bienia S, De Oliveira GS. Randomized equivalence trial of the King Vision aBlade videolaryngoscope with the Miller direct laryngoscope for routine tracheal intubation in children <2 yr of age. Br J Anaesth. 2017 Jun 1;118(6):932-937. doi: 10.1093/bja/aex073. PMID 28549081